CLINICAL TRIAL: NCT02596958
Title: Available - Avastin in Addition to Platinum-based Chemotherapy is Indicated for First-lime Treatment of Patients With Locally Advanced, Metastatic or Recurrent Non-small Lung Cancer Other Than Predominantly Squamous Cell Histology
Brief Title: Safety and Efficacy Study of Avastin in Locally Advanced Metastatic or Recurrent Non-small Lung Cancer (NSLC) Participants
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML21217
Record Dates: First submitted 2015-11-03; First posted 2015-11-04 (Estimated); Results first posted 2016-03-04 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Bevacizumab: Patients will receive six 3-weeks cycle of IV bevacizumab along with platinum-based chemotherapy, followed by maintenance therapy of bevacizumab until progression (approximately 7 months).
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — Six 3-weeks cycle of IV bevacizumab will be administered for approximately 7 months.
  Other Names: Avastin

SUMMARY:
The purpose of this non-interventional study is the collection and documentation of data on safety and efficacy of intravenous (IV) bevacizumab (Avastin) in addition to platinum-based chemotherapy for first-line treatment in participants with unresectable advanced, metastatic or recurrent non-small cell lung cancer (NSCLC) other than predominantly squamous cell histology with focus on adenocarcinoma and elderly patients in daily routine.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to (>=) 18 years
* Histologically confirmed predominantly non-squamous NSCLC that is unresectably advanced, metastatic or recurrent (with or without adenocarcinoma)
* No contraindications to Avastin® according to the current Summary of Product Characteristics (SmPC) for Avastin®
* Therapeutic decision for Avastin® as first line treatment in combination with platinum-based chemotherapy was taken individually and independent of the non-interventional trial.

Exclusion Criteria:

N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with unresectable advanced, metastatic or recurrent non-small cell lung cancer other than predominantly squamous cell and with or without adenocarcinoma histology will be selected.
Sampling Method: Non-Probability Sample
Enrollment: 996 (Actual)
Dates: Start 2007-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Goslar, Germany

REFERENCES:
- [Derived] Zahn MO, Linck D, Losem C, Gessner C, Metze H, Gaillard VE, Tessen HW. AVAiLABLE NIS - AVASTIN(R) in lung cancer treatment in routine oncology practice in Germany. BMC Cancer. 2019 May 10;19(1):433. doi: 10.1186/s12885-019-5618-0. PMID 31077164

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab: Participants received bevacizumab (Avastin) in addition to platinum based chemotherapy for up to 6 cycles (21-day cycles) followed by bevacizumab as a single agent until disease progression. The dose and administration schedule was at the discretion of the treating physician and as per the recommendations given in the current summary of product characteristics (SmPC).
Period: Overall Study
Arm/Group | Bevacizumab
Started | 996
Completed | 0
Not Completed | 996
Not completed — Serious Adverse Drug Reactions | 44
Not completed — Cancer Progression | 441
Not completed — Death From Cancer | 112
Not completed — Death From Other Cause | 33
Not completed — Refusal of Treatment/Poor Cooperation | 61
Not completed — Administrative Reasons/Other | 231
Not completed — Lost to Follow-up | 33
Not completed — Missing | 32
Not completed — Excluded Due to Second Line Treatment | 9

BASELINE CHARACTERISTICS:
Population: Analysis population was defined as all participants included in the observational study, regardless of whether they finished it or not. Nine hundred and ninety six (996) participants were documented but only 987 participants were included in the analysis population as 9 participants were excluded due to documented second line treatment.
Groups:
- Bevacizumab: Participants received bevacizumab (Avastin) in addition to platinum based chemotherapy for up to 6 cycles (21-day cycles) followed by bevacizumab as a single agent until disease progression. The dose and administration schedule was at the discretion of the treating physician and as per the recommendations given in the current SmPC.
Arm/Group | Bevacizumab
Number analyzed (Participants) | 987
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (9.8)
Sex/Gender, Customized [Number; unit: participants]
  Female | 396
  Male | 590
  Missing | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Drug Reactions (ADRs), Toxicities, Avastin-Related ADRs, and Serious ADRs
Description: ADRs were defined as any response to a drug which was noxious and unintended, and which occurred at dose normally used related to the pharmacological properties. Serious ADRs were defined as any untoward medical occurrence or effect that at any dose resulted in death or life-threatening conditions or required hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, congenital anomaly or birth defect or medically important condition. Toxicity was defined as an adverse event that had an attribution (the relationship to investigational agent) of possible, probable or definite. Avastin-related ADRs (an adverse event with a possible relationship or a relationship to the treatment with AVASTIN) were due to Avastin. ADRs includes serious as well as non-serious ADRs.
Time Frame: Up to 74 months
Population: Analysis population was defined as all participants included in the observational study, regardless of whether they finished it or not.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 987
percentage of participants
  ADRs | 88.6
  Toxicities | 88.2
  Avastin-related ADR | 27.0
  Serious ADR | 11.1

2. Secondary Outcome: Percentage of Participants Who Withdrew or Modified Treatment
Description: Percentage of participants who withdrew treatment or experienced at least 1 dose deviation in relation to the planned Avastin therapy were reported.
Time Frame: Up to 74 months
Population: Analysis population was defined as all participants included in the observational study, regardless of whether they finished it.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 987
percentage of participants | 8.8

3. Secondary Outcome: Number of Cycles of Systemic Therapy
Description: Number of cycles of systemic therapy was the mean number of cycles received by participants in combination therapy with Avastin and chemotherapy and with Avastin monotherapy (maintenance).
Time Frame: Up to 74 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cycles
Arm/Group | Bevacizumab
Number analyzed (Participants) | 987
cycles
  Total number of cycles | 7.6 (7.0)
  Number of cycles with combination therapy | 4.2 (1.8)
  Number of cycles with maintenance therapy | 3.4 (6.2)

4. Secondary Outcome: Percentage of Participants With Best Tumor Response Over Time
Description: Best tumor response (assessed as per clinical routine of the individual center) was categorized according to the following criteria at the investigator discretion: complete response (CR: commonly defined as disappearance of all target lesions, all non-target lesions, and no new lesion), partial response (PR: commonly defined as at least a 30 percent [%] decrease in the sum of the longest diameter [LD] of target lesions, no progression in non-target lesion, and no new lesion), stable disease (SD: commonly defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD], in addition to no new target lesions). PD: commonly defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started and not evaluable (NE).
Time Frame: Up to 74 months
Population: Analysis population was defined as all participants included in the observational study, regardless of whether they finished it. Here, number of participants analyzed = participants with non-missing tumor response data.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 976
percentage of participants
  CR | 2.3
  PR | 43.3
  SD | 29.4
  PD | 10.1
  NE | 14.9

5. Secondary Outcome: Percentage of Participants With Eastern Cooperative Group(ECOG) Performance Status Grades
Description: ECOG Performance Status measured on-therapy (time between first dose and last dose date with a 30-day lag) assessed participant's performance status on 5 point scale: 0 is equal to (=) fully active/able to carry on all pre-disease activities without restriction; 1=restricted in physically strenuous activity, ambulatory/able to carry out light or sedentary work; 2=ambulatory (greater than [>] 50% of waking hours [hrs]), capable of all self care, unable to carry out any work activities; 3=capable of only limited self care, confined to bed/chair >50% of waking hrs; 4=completely disabled, cannot carry on any self care, totally confined to bed/chair; 5=dead.
Time Frame: Up to 74 months
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 806
percentage of participants
  Grade 0 | 18.7
  Grade 1 | 50.1
  Grade 2 | 23.2
  Grade 3 | 6.2
  Grade 4 | 1.7

6. Secondary Outcome: Percentage of Participants With Disease Control
Description: Disease control was defined as having achieved CR (commonly defined as disappearance of all target lesions, all non-target lesions, and no new lesion), PR (commonly defined as at least a 30% decrease in the sum of the LD of target lesions, no progression in non-target lesion, and no new lesion), or SD (commonly defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, in addition to no new target lesions) during the course of observation which were assessed as per investigator discretion. PD: commonly defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started and NE.
Time Frame: Up to 74 months
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 976
percentage of participants | 75.0

7. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time (months) between the start of therapy and progression (unequivocal progression of existing non-target lesions) or death. Progression: at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started. PFS was estimated using Kaplan-Meier method.
Time Frame: Up to 74 months
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab
Number analyzed (Participants) | 941
months | 7.4 [7.1 to 8.4]

8. Secondary Outcome: Percentage of Participants Who Died
Time Frame: Up to 74 months
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 975
percentage of participants | 17.5

9. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time (months) between the start of therapy and the date of death.
Time Frame: Up to 74 months
Population: Analysis population was defined as all participants included in the observational study, regardless of whether they finished it. Here 'number of participants analyzed' = participants assessed for this outcome measure.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Bevacizumab
Number analyzed (Participants) | 975
months | 18.4 (0.5)

ADVERSE EVENTS:
Time Frame: Up to the end of study (median duration of 170.8 days)
Arm/Group | Bevacizumab
Serious Adverse Events (participants affected / at risk) | 110/987
Other Adverse Events (participants affected / at risk) | 851/987
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab (N=987)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 15
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Acquired tracheo-oesophageal fistula (Respiratory, thoracic and mediastinal disorders) | 1
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Oesophagobronchial fistula (Respiratory, thoracic and mediastinal disorders) | 1
Pleural fistula (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 15
Haemorrhage (Vascular disorders) | 1
Pneumonia (Infections and infestations) | 9
Sepsis (Infections and infestations) | 4
Peritonitis (Infections and infestations) | 3
Large intestine perforation (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 3
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 1
Large intestinal haemorrhage (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Death (General disorders) | 4
Leukopenia (Blood and lymphatic system disorders) | 5
Anaemia (Blood and lymphatic system disorders) | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 2
Pancytopenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Splenic infarction (Blood and lymphatic system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 3
Cerebral ischaemia (Nervous system disorders) | 1
Cardiac failure (Cardiac disorders) | 4
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Proteinuria (Renal and urinary disorders) | 3
Fistula (Musculoskeletal and connective tissue disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab (N=987)
Anaemia (Blood and lymphatic system disorders) | 594
Leukopenia (Blood and lymphatic system disorders) | 492
Neutropenia (Blood and lymphatic system disorders) | 311
Thrombocytopenia (Blood and lymphatic system disorders) | 307
Pain (General disorders) | 171
Pyrexia (General disorders) | 102
Chest pain (General disorders) | 66
Hypertension (Vascular disorders) | 134
Pain in extremity (Musculoskeletal and connective tissue disorders) | 68
Back pain (Musculoskeletal and connective tissue disorders) | 50
Peripheral sensory neuropathy (Nervous system disorders) | 111
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 99
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 61
Proteinuria (Renal and urinary disorders) | 56
Nausea (Gastrointestinal disorders) | 459
Vomiting (Gastrointestinal disorders) | 185
Diarrhoea (Gastrointestinal disorders) | 99

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.